CLINICAL TRIAL: NCT01651182
Title: Open Label, Non-Randomized, Study to Evaluate the Pharmacokinetics of Tranexamic Acid in Patients Undergoing Major Liver Resection
Brief Title: Tranexamic Acid Versus Placebo for Blood to Reduce Perioperative Bleeding Post-liver Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Toronto (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TXA Liver - PK
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Cancer; Tumour; Surgery
Keywords: Blood transfusion; Blood loss; Postoperative complications; Outcome
MeSH Terms: conditions — Neoplasms; Hemorrhage; Postoperative Complications | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care (Placebo Comparator): No tranexamic acid
  Interventions: Drug: No tranexamic acid
- Dose 1 (Experimental): 1 g bolus + 1 g infusion from induction over 8 hours
  Interventions: Drug: Tranexamic Acid
- Dose 2 (Experimental): 1 g bolus + 10 mg/kg/hr from induction until end of surgery
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: No tranexamic acid — Control
  Arms: Standard Care
Drug: Tranexamic Acid
  Other Names: Cyklokapron
  Arms: Dose 1; Dose 2

SUMMARY:
Tranexamic acid (TXA) is an antifibrinolytic agent that has been shown to reduce blood loss and blood transfusion requirements in the following patient populations: multisystem trauma, liver transplantation, cardiac surgery and spine surgery. Patients undergoing major liver resection are at risk of severe perioperative blood loss and may also benefit from perioperative TXA administration.

This open label, non-randomized study to evaluate the pharmacokinetic and pharmacodynamic properties of two well studied dosing regimens of TXA will provide guidance in determining the optimal TXA dosing regimen for patients undergoing major liver resection. Compelling evidence of the effectiveness of TXA comes from the large multicentred, multi-national CRASH-2 trial where TXA was administered as a 1 g bolus + 1 g infusion over 8 hours. In liver transplant surgery, the following dose regimen has been shown to have great effect:10 mg/kg/h from the start of surgery until 2 hours after reperfusion of the liver transplant.

Although TXA is not currently approved for use in patients undergoing major liver resection, Health Canada has allowed the use of tranexamic acid for use in this research study.

ELIGIBILITY:
Inclusion Criteria

* Patient undergoing anticipated open or laparoscopic major liver resection (> 2 hepatic segments), as assessed by the operating surgeon
* Age ≥ 18 years.

Exclusion Criteria

* Previously enrolled in this study
* Platelet count less than 100,000/mm3
* Severe anemia (hemoglobin levels less than 90 g/l)
* Documented arterial or venous thrombosis at screening or in past three months
* Anticoagulants (other than LMWH or heparin in prophylactic doses to prevent deep vein thrombosis), direct thrombin inhibitors or thrombolytic therapy administered or completed within last week
* Hepatectomy associated with planned vascular or biliary reconstruction
* Known disseminated intravascular coagulation
* Severe renal insufficiency (CrCl<30)
* History of seizure disorder
* Pregnant or lactating
* Hypersensitivity to tranexamic acid or any of the ingredients
* Unable to receive blood products (i.e. difficulty with cross matching, refuses blood transfusion, or a past history of unexplained severe transfusion reaction)
* Receipt of chemotherapy within 4 weeks of scheduled operation
* Patients undergoing resection for living donor liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Receipt of blood transfusion(s) | 7 days

SECONDARY OUTCOMES:
Fibrinolytic Markers | Baseline - Postoperative Day 0-7
Pharmacokinetic Study | Baseline - Postoperative Day 0-7
Post-operative incidence of symptomatic venous thromboembolic event | 30 days
Other post-operative complications | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Karanicolas PJ, Lin Y, Tarshis J, Law CH, Coburn NG, Hallet J, Nascimento B, Pawliszyn J, McCluskey SA. Major liver resection, systemic fibrinolytic activity, and the impact of tranexamic acid. HPB (Oxford). 2016 Dec;18(12):991-999. doi: 10.1016/j.hpb.2016.09.005. Epub 2016 Oct 18. PMID 27765582